CLINICAL TRIAL: NCT01932502
Title: Evaluation of Onfi Conversion Therapy Replacing Clonazepam in Patients With Medically Refractory Epilepsy: Efficacy, Tolerability, Dosing Equivalence, and Retention Rate
Brief Title: Evaluation of Onfi Conversion Therapy Replacing Clonazepam in Patients With Medically Refractory Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13BN001
Record Dates: First submitted 2013-08-23; First posted 2013-08-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Refractory Epilepsy
Keywords: epilepsy; Onfi; clonazepam
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — Clobazam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clonazepam conversion to clobazam (Onfi) (Experimental): Subject's clonazepam will be converted to clobazam (Onfi). This is an open label study without placebo control.
  Interventions: Drug: clobazam (Onfi); Drug: Initial conversion and titration; Drug: Conversion schedule - Week 1; Drug: Conversion schedule - Week 2; Drug: Conversion schedule - Week 3

INTERVENTIONS:
Drug: clobazam (Onfi) — Subject's clonazepam will be converted to the following Onfi doses per day:
  Clonazepam 0.5mg converted to Onfi 10mg first week, then titrated up to 40mg per day.
  Clonazepam 1.0-2.0mg converted to Onfi 20mg first week, then titrated up to 40mg per day.
  Clonazepam 2-4mg converted to Onfi 20mg first week, then titrated up to 60mg per day.
  Initial conversion will occur over two weeks followed by upward titration of up to 10mg increment per week toward the target dose. Down titration of up to 10mg will be allowed during the study.
  The following will be the initial conversion schedule from clonazepam to Onfi:
  Week 1: 50% reduction of clonazepam and starting dose of Onfi, replacing the reduced clonazepam dose with the conversion rate of clonazepam 0.5mg = Onfi 10mg.
  Week 2: Discontinuing clonazepam and increasing the dosage of Onfi by two-fold. Week 3+: Titrate the dose of Onfi up to 40mg per day as tolerated
Drug: Initial conversion and titration — Initial conversion will occur over two weeks followed by upward titration of up to 10mg increment per week toward the target dose. Down titration of up to 10mg will be allowed during the study.
  Other Names: clobazam (Onfi)
Drug: Conversion schedule - Week 1 — The following will be the initial conversion schedule from clonazepam to Onfi:
  Week 1: 50% reduction of clonazepam and starting dose of Onfi, replacing the reduced clonazepam dose with the conversion rate of clonazepam 0.5mg=Onfi 10mg.
  Other Names: clobazam (Onfi)
Drug: Conversion schedule - Week 2 — Week 2: Discontinuing clonazepam and increasing the dosage of Onfi by two-fold.
  Other Names: clobazam (Onfi)
Drug: Conversion schedule - Week 3 — Week 3+: Titrate the dose of Onfi up to 40mg per day as tolerated.
  Other Names: clobazam (Onfi)

SUMMARY:
The purpose of the study is to examine the clinical safety, tolerability, and efficacy of clobazam (Onfi) when it replaces the pre-existing clonazepam therapy in patients with refractory epilepsy.

DETAILED DESCRIPTION:
The study is designed to answer frequently asked questions when clinicians replace existing 1,4-benzodiazepine to Onfi, as follows:

1. What should be the optimal equivalent doses for conversion?
2. How quickly should it be converted?
3. Would there be significant improvement of seizure control?
4. Should we expect difference in tolerability? If so, what are common adverse events?
5. Would the tolerance to the therapeutic effect differ with Onfi after conversion?

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of medically refractory epilepsy with or without secondary generalization for at least 12 months prior to the initial study visit.
* Currently taking stable dosing regimen of clonazepam (0.5-4mg daily) for seizure control.
* Takes at least one additional Anti-epileptic drug besides benzodiazepine.
* Age 18-70 years, inclusive.
* In opinion of investigator, can be safely treated with Onfi.
* Minimum of 2 seizures, but no more than 24 complex partial or generalized seizures, during the 8-week baseline period prior to study entry.
* Able to communicate effectively with study personnel and considered reliable, able, willing, and cooperative with regard to complying with protocol-defined requirements, including completion of study diary.

Exclusion Criteria:

* Clinically relevant current illness or history of that may interfere with the subject's ability to complete the study as determined by the investigator.
* History of status epilepticus within 6 months prior to the initial study visit.
* History of suicidal attempts or suicidal ideation within 12 months of initial visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 28 days
  Efficacy will be measured by percentage of mean seizure reduction averaged over 28 days.

SECONDARY OUTCOMES:
Tolerability | Weeks 6 - 52 after medication conversion
  Retention rate, which indirectly measures the therapeutic tolerance, will be measured at 6 weeks, 12 weeks, 24 weeks, and 52 weeks.
Retention | 52 weeks
  Retention rate of Onfi at 6-months and 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Chung, MD, Principal Investigator — Banner Health Systems
Locations (1):
- Banner Health, Phoenix, Arizona, United States